CLINICAL TRIAL: NCT05646147
Title: Diagnostic Accuracy of the Maximal Systolic Acceleration for Detection of Peripheral Arterial
Brief Title: DIAbetes Maximal ACCeleration
Acronym: DIAMACC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, jjwmbrouwers, Surgical Resident, MD, PhD-candidate, post-doc, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LUMC-DIAMACC
Record Dates: First submitted 2022-11-20; First posted 2022-12-12 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Peripheral Arterial Disease; Diagnosis; Diabetic Foot
Keywords: Peripheral Arterial Disease; Diabetic Foot; Diagnosis
MeSH Terms: conditions — Peripheral Arterial Disease; Disease; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic Cohort Study (Other): All patients will underwent full diagnostic testing.
  Interventions: Device: Maximal Systolic Acceleration

INTERVENTIONS:
Device: Maximal Systolic Acceleration — Reliability of the maximal systolic acceleration

SUMMARY:
Prevalence of diabetes mellitus (DM) is increasing rapidly, with patient numbers projected to rise to 643 million by 2030. As a consequence of diabetes-related atherosclerosis, peripheral arterial disease (PAD) and in particular medial arterial calcification (MAC) can occur. The accurate identification of PAD by bedside tests is extremely important in patients with diabetes and foot ulceration, in order to reduce delayed wound healing, prevent lower limb amputation and eventually reduce mortality. However, as shown in previous systematic reviews, the performance of current bedside tests is not reliable in excluding PAD in diabetic patients.1,2 Moreover, the methodological quality of the conducted studies is generally poor. Therefore, more reliable and prospective data is required. Also alternative bedside tests need to be investigated. As an example, the ACCmax (a new doppler derived parameter) could be particularly promising in this patient group.

DETAILED DESCRIPTION:
According to the latest 2021 data from the International Diabetes Federation, an estimated 537 million adults are living with DM globally.3 Prevalence is increasing rapidly, with numbers projected to rise to 643 million by 2030 and 783 million by 2045. Annually, DM causes 6.7 million deaths, as a consequence of both macrovascular- (atherosclerosis) and microvascular disease (retinopathy, nephropathy, and neuropathy). In 2021, diabetes caused at least 966 billion dollars in health expenditure, comprising approximately 9% of total spending on adults. Type 2 diabetes comprises about 85-90% of these cases, in which disease onset is often insidious, and diagnosis is consequently delayed.4

Peripheral arterial disease (PAD) of the lower extremity is a clinical manifestation of systemic atherosclerosis and considered a well-known (long-term) complication of DM. Besides atherosclerosis, calcification of the tunica media of the arterial wall can occur. This process is called medial arterial calcification (MAC) and is accelerated in the presence of DM. Research suggests that MAC is present in approximately one third of patients with DM.5 MAC has been shown to be an independent predictor of cardiovascular mortality, while another study found that patients with DM and PAD have an impaired quality of life and an increased risk of adverse cardiac and limb events.6,7

Timely recognition of limb ischemia is important in patients with DM/MAC in order to reduce delayed wound healing, prevent lower limb amputation and eventually reduce mortality.8 Current non-invasive bedside tests - such as the ankle-brachial index (ABI) and toe pressure (TP) - are considered accurate for the diagnosis of PAD. However, as shown in previous systematic reviews, the performance of current bedside tests is not reliable in excluding PAD in diabetic patients.1,2 The methodological quality of the studies in these reviews were poor. In general, most of the data was collected retrospectively and not all patients received reference testing. In order to assess the reliability of bedside tests in this patient group, more well-sound methodological research is required. Also alternative bedside tests need to be investigated.

The doppler derived maximal systolic acceleration (ACCmax) is a new non-invasive parameter, which could be promising in detecting PAD. Although ACCmax has already been used for renal artery stenosis9, thorough evaluation has not been performed in PAD. Two previous studies showed accurate diagnostic property in diabetic patients, but the sample sizes were small.10,11

The aim of this study is to assess the clinical value of bedside tests compared to DUS to detect PAD in patients with diabetes-related foot ulceration, with special emphasis on the ACCmax.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* DM in medical history.
* Presenting with a new-onset wound or ulceration on the foot or ankle with initiation of a new diagnostic care path.

Exclusion Criteria:

- Lacking capacity to consent for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Reliability of standard bedside tests and the maximal systolic acceleration (ACCmax) | Through study completion, approximately 1.5 years
  Sensitivity and specificity including their derivates: PLR and NLR

SECONDARY OUTCOMES:
Comparison of ACCmax reliability with current bedside tests | Through study completion, approximately 1.5 years
  Comparison of ACCmax reliability with current bedside tests
Comparison of patient demographics (such as age/sex) and comorbidities (duration of diabetes, chronic kidney disease) with diagnostic accuracy of different bedside tests | Through study completion, approximately 1.5 years
  Comparison of patient demographics (such as age/sex) and comorbidities (duration of diabetes, chronic kidney disease) with diagnostic accuracy of different bedside tests
Wound healing and ACCmax | Up to 5 years after study completion
  To assess if the maximal systolic acceleration can predict wound healing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Willems S, Schepers A, Hamming J, Brouwers JJWM. DIAMACC: protocol of a prospective diagnostic accuracy study of the maximal systolic acceleration to detect peripheral arterial disease in patients with diabetes-related foot ulceration in the Netherlands. BMJ Open. 2024 Dec 20;14(12):e086629. doi: 10.1136/bmjopen-2024-086629. PMID 39806662